CLINICAL TRIAL: NCT00215241
Title: Placebo-Controlled Trial of Risperidone Augmentation for SSRI-Resistant Civilian PTSD
Brief Title: Risperidone Augmentation for PTSD
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Janssen Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5816; 5816-05-4R1 (Other: Duke legacy protocol ID)
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2014-09-22 (Estimated); Status verified 2006-06

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: PTSD; sertraline; risperidone; antidepressant; antipsychotic; anxiety; trauma
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Anxiety Disorders; Wounds and Injuries | interventions — Sertraline; Risperidone

INTERVENTIONS:
Drug: sertraline and risperidone

SUMMARY:
The purpose of this study is to (1) compare the response of civilians with Posttraumatic Stress Disorder(PTSD) currently receiving sertraline without an optimal response to risperidone augmentation vs. placebo, and (2) to evaluate the tolerability of risperidone augmentation, and (3) to identifiy predictors of response to risperidone augmentation. the hypothesis is that risperidone augmentation of sertraline treatment of PTSD is safe and effective.

DETAILED DESCRIPTION:
This is a multi-center, two-phase study to evaluate the efficacy and safety of risperidone augmentation to sertraline treatment of Post-Traumatic Stress Disorder (PTSD). In the first phase, all patients will be assigned to take open label sertraline for 8 weeks (up to 200 mg/d). Those who have not achieved a significant decrease in their PTSD symptoms by week 8 will be entered into the second phase. In the second phase, patients will continue with the sertraline, but will then be randomly given either risperidone (up to 3 mg/d) or matching placebo in double-blind fashion.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent prior to any study procedures being done
* Male or female outpatients between 18-65 years of age
* Trauma experienced meets trauma defined by DSM
* Meets criteria for DSM-IV PTSD as a result of civilian trauma
* CAPS Score of greater than or equal to 50 at screening and baseline
* Able to swallow whole capsules
* Fluency in both written and spoken English
* Negative urine drug screen at screening visit
* If female of childbearing potential, must have negative serum pregnancy test at screening visit and must agree to use a medically accepted means of contraception throughout the study and for 30 days after completion of the study
* To be include in Phase 2, must complete Phase I and must have less than 70% reduction from baseline on the CAPS

Exclusion Criteria:

* Pregnant women or those likely to become pregnant, or nursing mothers
* Medical instability (clinically significant hepatic, cardiac, or pulmonary disease, HIV, uncontrolled hypertension, diabetes or thyroid conditions, seizure disorders, clinically significant laboratory abnormalities at screen
* Primary psychotic disorder, or history of schizophrenia, other psychotic disorder, bipolar disorder, or cognitive disorder
* Those considered a risk for suicidal or homicidal behavior (the clinician will immediately, upon assessing a risk for suicidal or homicidal behavior, refer the patient for further evaluation and probable hospitalization)
* Hypersensitivity or other contraindication to sertraline or risperidone
* Meeting DSM-IV criteria for drug or alcohol dependence within 3 months of study entry
* Those who are still experiencing an ongoing traumatic stressor (domestic violence/elder abuse) who will need to focus on safety (the clinician will make referrals as appropriate)
* DSM-IV primary diagnosis of any other anxiety disorder or major depressive disorder
* Current use of antipsychotic, or other psychotropic medications, or supplements with known psychotropic effects
* Current involvement in litigation related to PTSD
* Current psychotherapy aimed at treating PTSD
* PTSD as a result of combat-related trauma
* Previous failure to respond to sertraline-risperidone combination at therapeutic dose

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2004-04; Study Completion 2006-07

PRIMARY OUTCOMES:
Clinician Administered PTSD Scale (CAPS)

SECONDARY OUTCOMES:
Davidson Trauma Scale (DTS)
Beck Depression Inventory
Quality of Life/Q-LES-Q
Connor-Davidson Resilience Scale
Clinical Global Improvement Scale (CGI-I)
Positive and Negative Symptoms Scale (PANSS)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Davidson, M.D., Principal Investigator — Duke University; Barbara Rothbaum, Ph.D., Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University Medical Center, Atlanta, Georgia
  - Medical University of South Carolina, Charleston, South Carolina